CLINICAL TRIAL: NCT05323812
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Pharmacodynamics and Pharmacokinetics of TW001 in Alzheimer Patients
Brief Title: ASURE: Alzheimer Study Using oRal Edaravone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Treeway B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TW001-AD-C2.01; 2021-003164-27 (EudraCT Number)
Record Dates: First submitted 2022-03-16; First posted 2022-04-12 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Oxidative stress biomarkers; Free radical scavenger; Edaravone
MeSH Terms: conditions — Alzheimer Disease | interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- TW001 (Experimental)
  Interventions: Drug: TW001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TW001 — daily dose of 100 mg TW001/placebo
  Other Names: Edaravone
  Arms: TW001
Drug: Placebo — daily dose of 100 mg TW001/placebo
  Arms: Placebo

SUMMARY:
This is a multi-center, Phase IIa, randomized, double-blind, placebo-controlled study in patients with Alzheimer's Disease (AD).

DETAILED DESCRIPTION:
This is an exploratory, double-blind, randomized, placebo-controlled phase IIa proof of concept study to evaluate the safety, pharmacodynamics and pharmacokinetics of TW001 in patients with mild AD. Patients will be randomized 1:1 to TW001 and placebo. Treatments will be given in a fasted state once daily for 90 days. The total duration of the clinical trial will be approximately 4 months per patient.

ELIGIBILITY:
Inclusion Criteria:

1. Age 55-80 years (both inclusive), male or female.
2. Body mass index between 18.5 to 33.0 kg/m2 (both inclusive).
3. Should meet the criteria for early clinical stage Alzheimer's Disease (AD) according to the National Institute on Aging and Alzheimer's Association (NIA-AA) criteria research framework:

   1. Gradual and progressive change in memory function reported by patient or informant over more than 6 months,
   2. Clinical syndrome of Mild Cognitive Impairment (MCI) due to AD or mild AD dementia,
   3. An Mini-Mental State Exam (MMSE) score ≥ 20 at screening,
   4. Biomarker classification according to the Amyloid/Tau/Neurodegeneration (ATN) as A+T+N+ or A+T+N- based upon:

   (i) Cerebrospinal fluid (CSF) profile consistent with AD (an Aβ42 concentration of <1000 pg/mL AND phosphorylated tau (p-tau) >19 pg/mL, or a ratio of p-tau/Aβ42 of ≥0.020) taken during the screening period prior to the day of the first dose of study medication, or

   (ii) Documented evidence of a CSF profile consistent with AD obtained with the previous 12 months, or

   (iii) Documented amyloid positron emission tomography (PET) scan evidence acquired within the previous 12 months.
4. A reliable and competent trial partner/caregiver who can assist and witness dosing and is willing to accompany the patient to all visits. The trial partner/caregiver should understand the nature of the trial and adhere to trial requirements (e.g., visit schedules, evaluations) and confirm this by co-signing the informed consent of the patient or signing of a separate informed consent of the partner/caregiver according to the local requirements.
5. If a patient is taking medication, supplements or vitamins that may have an influence on oxidative stress, cognition and/or EEG, the dose must be stable at screening for at least one month, and the patient must be willing to remain on the same treatment and dose for the duration of the trial.
6. A male patient abstains from sexual intercourse, or is vasectomized (> 6 months), or will use a condom with spermicide during sexual intercourse during the trial and for three months after participation in the trial and will abstain from sperm donation during the trial and for three months after participation in the trial.
7. A female patient should not be of reproductive potential:

   A female patient who is not of reproductive potential is defined as one who:
   1. Has reached natural menopause (defined as 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone [FSH] levels in the postmenopausal range as determined by the local laboratory, or 12 months of spontaneous amenorrhea);
   2. Is 6 weeks post-surgical bilateral oophorectomy with or without hysterectomy; or
   3. Has undergone bilateral tubal ligation. Spontaneous amenorrhea does not include cases for which there is an underlying disease that causes amenorrhea (e.g., anorexia nervosa).
8. Capable of providing informed consent and complying with trial procedures.

Exclusion Criteria:

1. A known history of stroke that is clinically important in the investigator's opinion.
2. Evidence of a clinically relevant neurological disorder other than AD at screening, including but not limited to: vascular dementia, Parkinson's disease, frontotemporal dementia, Huntington's disease, amyotrophic lateral sclerosis, multiple sclerosis, progressive supranuclear palsy, dementia with Lewy bodies, other types of dementia, neurosyphilis or head trauma with loss of consciousness that led to persistent cognitive deficits.
3. A history of seizures or epilepsy within the last 5 years before screening.
4. Evidence of a clinically relevant or unstable psychiatric disorder, based on the 5th edition after text revision of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5TM) criteria, including schizophrenia or other psychotic disorder, bipolar disorder, major depression, or delirium. Major depression in remission is not exclusionary.
5. Renal impairment as indicated by a creatinine clearance of less than 50 mL/min as calculated by the Cockcroft Gault equation.
6. Patient has a history of any of the following conditions:

   1. Clinically significant hepatic disease,
   2. AST or ALT levels of ≥ 2 times upper limit of normal (ULN),
   3. Biliary tract disease,
   4. Patient has a positive screening test for HIV, hepatitis B or C.
7. Presence of any of the following clinical conditions:

   1. Unstable cardiac, pulmonary, endocrine, hematologic or active infectious disease,
   2. Unstable psychiatric illness defined as psychosis, untreated major depression within 90 days of the screening visit,
   3. A history of cancer within the past 3 years prior to screening other than treated squamous cell carcinoma, basal cell carcinoma and melanoma in situ, or in-situ prostate cancer or in-situ breast cancer which have been fully removed and are considered cured
8. History or signs/symptoms of lumbar spine/disc disease including but not limited to scoliosis, herniation, or any other contraindication to lumbar puncture.
9. History of known sensitivity or intolerability to edaravone, related substances of edaravone, or to any of the excipients.
10. Current substance or alcohol dependence.
11. Exposure to any investigational drug within 30 days of the screening visit.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Nature, frequency and severity of adverse events | Through study completion, up to 4 months
  Safety and tolerability as measured by nature, frequency and severity of adverse events and serious adverse events
Plasma oxidative stress biomarkers | Through study completion, up to 4 months
  Changes from baseline in: 8-OHdG/8-OHG and Uric acid in plasma
Cerebrospinal Fluid (CSF) oxidative stress biomarkers | Through study completion, up to 4 months
  Changes from baseline in: 8-OHdG/8-OHG in CSF

SECONDARY OUTCOMES:
Plasma concentration of TW001 | Through study completion, up to 4 months
Area under the concentration versus time curve (AUC) of TW001 | Through study completion, up to 4 months
Maximum plasma concentration (Cmax) of TW001 | Through study completion, up to 4 months
Time to reach maximum plasma concentration (tmax) of TW001 | Through study completion, up to 4 months

OTHER OUTCOMES:
Plasma biomarkers of AD pathology and neurodegeneration | Through study completion, up to 4 months
  Changes from baseline in: Aβ42, Aβ40, phosphorylated tau epitopes, GFAP and NfL
CSF biomarkers of AD pathology and neurodegeneration | Through study completion, up to 4 months
  Changes from baseline in: Aβ42, Aβ40, phosphorylated tau epitopes, t-tau, GFAP, YKL-40, NfL and NRGN
Urine oxidative stress biomarkers | Through study completion, up to 4 months
  Changes from baseline in: 8-OHdG/8-OHG in urine
Cognitive assessment - Clinical Dementia Rating - Sum of Boxes (CDR-SB) | Through study completion, up to 4 months
  Change from baseline in CDR-SB score

CONTACTS AND LOCATIONS:
Locations (6):
- Croatia (2):
  - University Hospital Centre Osijek, Osijek
  - University Hospital Centre Zagreb, Zagreb
- Netherlands (4):
  - Brain Research Center Den Bosch, 's-Hertogenbosch
  - Brain Research Center Amsterdam, Amsterdam
  - ETZ Elisabeth ziekenhuis, Tilburg
  - Brain Research Center Zwolle, Zwolle

IPD SHARING:
Plan to Share IPD: No